CLINICAL TRIAL: NCT07351929
Title: An Emotional-distress-based Integrated Care Programme in Patients With an Acute Exacerbation of COPD (EmoD) - A Feasibility Study
Brief Title: Emotional-distress-based Integrated Care Programme in Patients With an Acute Exacerbation of COPD
Acronym: EmoD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-01178
Record Dates: First submitted 2025-11-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: COPD Exacerbation
Keywords: COPD; Feasibility study; Mixed-methods design; Emotional distress; Integrated care programme; APN
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Explanatory sequential mixed-methods design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Other: EmoD Intervention

INTERVENTIONS:
Other: EmoD Intervention — Patients who are hospitalised due to a COPD exacerbation will be aligned to a nurse-led emotional-distress-based integrated care programme for three months.

SUMMARY:
The investigators have developed a new counseling service that focuses on the emotional distress experienced by people living with COPD. The service has been specially developed for patients who have experienced a deterioration in their lung condition (known as an acute exacerbation of COPD). The new program is led by an APN team. Other professionals are involved in the program, such as medical staff and physiotherapists. The new counseling service lasts three months. Patients will receive ten counseling sessions with a specialized nurse.

The overall objective of the study is to assess the feasibility of the newly developed emotional-distress-based integrated care programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of COPD (GOLD 1-4)
* Hospitalisation due to a COPD exacerbation and decision to start with steroids and/or antibiotics (severe exacerbation)
* Age ≥ 18
* Inpatient on the pneumology or medical ward

Exclusion Criteria:

* Cognitive impairment (dementia, delirium) (DOS>3 or AES>6 or Mini-Cog<3)
* Unstable psychiatric disorders
* Not speaking German
* Lung transplant
* Pneumonia caused by chronic colonization by bacteria (Legionella, nontuberculous mycobacteria (NTM))
* Unable to telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in COPD-related emotional distress (CRED) | Quantitative data will be collected baseline, in the first month after hospitalization due to AECPOD (MZP 1, week 0-4), and follow-up, three months after (MZP2, week 14-17)
  Change in COPD-related emotional distress between baseline and month 3. COPD-related emotional distress will be assessed using the newly developed 'COPD-Related Emotional Distress Questionnaire (CRED)', which was developed for CF and COPD patients (publication in progress; former name of the questionnaire: IRED-RESP). The questionnaire includes 36 items and assesses distress related to symptoms, treatment, restrictions in range of mobility and participation in social life, unpredictability of the disease, and stigma, using a 5-point Likert scale. Higher scores mean more emotional distress (worse outcome).

SECONDARY OUTCOMES:
Reach: Total number of patients who take up the programme | Four months
  Number of patients who accept the study and / or intervention is documented by the study team.
Reach: Percentage of patients who take part in at least one outpatient intervention | Four months
  Number of interventions per patient and number of patients with termination of the programme before Week 13 is documented by the ANP team
Reach: Reasons for participating in the programme (facilitators and barriers) | Four months
  Patients who decline the intervention are asked by the ANP team and/or the study nurse for their reasons (barriers). The reasons for taking up the programme (facilitators) will be qualitatively investigated in interviews. A semi-structured interview guide will be used.
Reach: Reasons for ending (prematurely or on schedule) the programme (facilitators and barriers) | Four months
  The reasons for ending (prematurely or on schedule) the programme will be qualitatively investigated in interviews. A semi-structured interview guide will be used.
Potential effectiveness: Change in depression | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Depression will be screened with the Hospital Anxiety and Depression Scale (HADS). The concept is measured with seven 4-point rating scales ranging from 0 to 3. The sum score ranging from 0 to 21 will be calculated (Zigmond & Snaith, 1983). Higher scores meaning worse outcomes. Differences between MZP1 and MZP2 will be calculated per subscore.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in anxiety | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Anxiety will be screened with the Hospital Anxiety and Depression Scale (HADS). The concept is measured with seven 4-point rating scales ranging from 0 to 3. The sum score ranging from 0 to 21 will be calculated (Zigmond & Snaith, 1983). Higher scores meaning worse outcomes. Differences between MZP1 and MZP2 will be calculated per subscore.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health-related quality of life (QoL) | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Health-related quality of life will be assessed with the Chronic Respiratory Questionnaire (CRQ) (Guyatt et al., 1987) following the defined procedure of the developers. The self-administered questionnaire version with standardised dyspnea questions (SAS) will be used. The questionnaire was developed for patients with chronic airflow limitations and comprises 20 items which assess four domains: 1) dyspnea, 2) fatigue, 3) emotional function and 4) mastery. The scoring scale ranges from 1 (extreme) to 7 (not at all) and will be assessed with a recall period of the past two weeks. A subscore for each domain (sum of items / number of items) will be calculated. The CRQ-SAS is available in German. It has demonstrated high sensitivity in the evaluation of a rehabilitation programme (Puhan et al., 2007). Differences between MZP1 and MZP2 will be calculated per subscore.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Patient satisfaction with programme | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative The questionnaire on the quality of nursing care counseling (ANP-BQ) is used to assess patient satisfaction. This instrument includes, for example, a question to assess the satisfaction of care provided by the ANP on an NRS 1-10 (Petry et al., 2014; Weilenmann et al., 2021).
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Number of moderate exacerbations within 3 months | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative The number of moderate exacerbations during the previous three months are assessed at week 14-17. For this purpose, moderate exacerbations are defined as an acute (more than normal day-to-day variation) worsening of respiratory symptoms (breathlessness, sputum and / or coughing) that are treated with systemic antibiotics and / or corticosteroids (systemic = oral or intravenous) (Global Initiative for Chronic Obstructive Lung Disease, 2019).
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Number of severe exacerbations within 3 months | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative The number of severe exacerbations during the previous three months are assessed at week 14-17. For this purpose, severe exacerbations are defined as acute (more than normal day-to-day variation) worsening of respiratory symptoms (breathlessness, sputum and / or coughing) that result in hospitalisation or emergency room visit (Global Initiative for Chronic Obstructive Lung Disease, 2019).
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Rehospitalisation at day 90 | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative The number of COPD-related rehospitalisations after 3 months is assessed by medical chart review.
  Qualitative In the case of rehospitalisation, a one-to-one interview and medical chart review will be performed to assess reasons for rehospitalisation.
Potential effectiveness: Time until first rehospitalisation | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative The time until first rehospitalisation is assessed by medical chart review.
  Qualitative In the case of rehospitalisation, a one-to-one interview and medical chart review will be performed to assess reasons for rehospitalisation.
Potential effectiveness: Change in health behaviour smoking- current status | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Smoking behaviour will be assessed by using the questionnaire from the WHO (Global Adult Tobacco Survey Collaborative Group, 2011). It assesses the current status of smoking (yes / no).
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour smoking - ex- smoker | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Smoking behaviour will be assessed by using the questionnaire from the WHO (Global Adult Tobacco Survey Collaborative Group, 2011). If an ex-smoker, it assesses date of smoking cessation (year).
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour smoking -smoker | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Smoking behaviour will be assessed by using the questionnaire from the WHO (Global Adult Tobacco Survey Collaborative Group, 2011). If a smoker, it assesses the substance and the number per day.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour nutrition - body weight | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Current body weight (kg) will be assessed.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour nutrition - body height | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Current body height (m) will be assessed.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour nutrition - BMI | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Current Body Mass Index (BMI) will be calculated according to the WHO recommendations (World Health Organization, 2000) (kg/m^2).
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour nutrition - NRS | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Current Nutritional Risk Screening (NRS) will be assessed during hospitalisation (Kondrup et al., 2003). 3 and more points meaning worse outcome.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour physical activity - C-PPAC | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Self-report by patient based on the first two items of the clinical version of PROactive Physical Activity in COPD instrument (C-PPAC). The items measure the amount of activity over the last 7 days with a range from 0-4. Higher scores meaning better outcomes.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour physical activity - PR | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative The use of pulmonary rehabilitation/outpatient physiotherapy is recorded.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour inhalation adherence | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Adherence to inhalation will be assessed. The items were derived from the Zurich Assessment of Therapy Adherence CF (ZATA-CF) and adapted slightly. Patients are asked how often they needed to inhale the medication per day and how often they had skipped an inhalation in the past seven days. Higher scores meaning worse outcomes.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour action plan | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Availability of a prescription for an action plan (with/without self-medication) and adherence of patient to the action plan will be assessed.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Potential effectiveness: Change in health behaviour oxygen use | Study duration per patient is three months with two measurement points. Baseline measurement (MZP1) will be applied in the first month after hospitalization due to AECPOD (week 0-4). Second measurement (MZP 2) will take place in month four (week 14-17).
  Quantitative Availability of an oxygen prescription and the patient's compliance with the prescription are assessed.
  Qualitative A semi-structured interview guide will be used based on the quantitative results.
Implementation: Percent of programme components carried out according to the intervention manual | Data will be collected at the earliest six months after the start of the programme
  Quantitative Completed intervention components per patient were documented by the ANP team. Necessary but not or not fully completed parts of the intervention are also documented.
  Qualitative To understand reasons for performing, omitting or modifying components of the programme structured small group interviews will be conducted with HCP's involved in intervention delivery. The interview guide will be based on the results of the document analysis.
Implementation: Acceptability of the programme | Data will be collected at the earliest six months after the start of the programme
  Quantitative The German translations of the Acceptability of Intervention Measure (AIM) scale will be used to assess the healthcare professional's perspective. The scale contains four items; all are rated on a 5-point response scale (1 = completely disagree, 5 = completely agree), we added a sixth option "no response" (0 points).
  Qualitative To understand reasons for the results structured small group interviews will be conducted with involved HCPs. The interview guide will be based on the results of the questionnaires.
Implementation: Appropriateness of the programme | Data will be collected at the earliest six months after the start of the programme
  Quantitative The German translations of the Intervention Appropriateness Measure (IAM) scale will be used to assess the healthcare professional's perspective. The scale contains four items; all are rated on a 5-point response scale (1 = completely disagree, 5 = completely agree), we added a sixth option "no response" (0 points).
  Qualitative To understand reasons for the results structured small group interviews will be conducted with involved HCPs. The interview guide will be based on the results of the questionnaires.
Implementation: Feasibility of the programme | Data will be collected at the earliest six months after the start of the programme
  Quantitative The German translations of the Feasibility of Intervention Measure (FIM) scale will be used to assess the healthcare professional's perspective. The scale contains four items; all are rated on a 5-point response scale (1 = completely disagree, 5 = completely agree), we added a sixth option "no response" (0 points).
  Qualitative To understand reasons for the results structured small group interviews will be conducted with involved HCPs. The interview guide will be based on the results of the questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No